CLINICAL TRIAL: NCT02780765
Title: Study to Compare the Effect of Two Different Types of Humidifier on the Endotracheal Tube Patency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Vijaya P Patil, professor and Anaesthetist, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1665
Record Dates: First submitted 2016-05-11; First posted 2016-05-23 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Cancer of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heated humidifier group (Experimental): 30 postoperative patients with overnight endotracheal intubation will be supplied humidified oxygen using Heated Humidifier (HH). Temperature of inspired gas at the Y piece will be measured as surrogate marker for quality of humidification. The suctioning of ETT will be done once every 2 hourly by nurse/ doctor/trained personnel.
  Interventions: Device: heated humidifier
- Mist humidifier group (Active Comparator): 30 postoperative patients with overnight endotracheal intubation will be supplied humidified oxygen using mist nebuliser. Temperature of inspired gas at the Y piece will be measured as surrogate marker for quality of humidification. The suctioning of ETT will be done once every 2 hourly by nurse/ doctor/trained personnel.
  Interventions: Device: mist humidifier

INTERVENTIONS:
Device: heated humidifier — 30 patients requiring overnight intubation but breathing spontaneously without ventilatory support will be supplied humidified oxygen using Heated Humidifier(HH)
  Arms: Heated humidifier group
Device: mist humidifier — 30 patients requiring overnight intubation but breathing spontaneously without ventilatory support will be supplied humidified oxygen using mist humidifier
  Arms: Mist humidifier group

SUMMARY:
60 post operative patients who are kept intubated overnight & are spontaneously breathing will be either supplied humidified oxygen Heated Humidifier(HH) or conventional mist nebulizer.

Temperature of inspired gas at the Y piece will be measured.

Sterile water will be used for HH & Mist nebuliser.

The suctioning of endotracheal tube (ETT) will be done once every 2 hourly by nurse/ doctor/trained personnel and additional suctioning if required.

DETAILED DESCRIPTION:
60 post operative patients who are kept intubated overnight & are spontaneously breathing will be selected in Tata Memorial Hospital (TMH), Mumbai. 30 patients will be supplied through humidified oxygen using FISHER & PAYKEL MR 370 Heated Humidifier(HH) & 30 patients through conventional mist nebulizer.

Temperature of inspired gas at the Y piece will be measured as surrogate marker for quality of humidification. Continuous monitoring of temperature will be done using standard monitor.

The reusable HH will be subjected to disinfection between patients. Sterile water will be used for HH & Mist nebuliser.

The suctioning of endotracheal tube (ETT) will be done once every 2 hourly by nurse/ doctor/trained personnel.

Based on patient's clinical condition , additional suctioning will be done. Frequency of additional suctioning , reason for suctioning will be noted.

Information regarding the age, sex, type of surgery of the patient, co-morbidity if any size of ETT, the time of commencement of humidification , duration of use of humidifier, time of extubation, any complication leading to discontinuation of humidifier, frequency of refilling of nebulizer chamber, volume of ETT before intubation etc. will be noted.

The amount of Endotracheal tube blockade caused by secretion will be measured immediately following extubation.

The volume of Endotracheal tube secretion / amount of blockade will be assessed by the following process-

* The bevel end & Murphy's eye of the Endotracheal tube will be sealed using sterile insulating tape so that it become water tight. The tube will be gradually filled with measured amount of sterile fluid using small volume syringe to increase the accuracy of measurement. The amount of fluid it can hold will be measured & noted.
* The volume of extubated tube will be measured in the similar way.
* The measured volume of the Extubated Endotracheal tube will be subtracted from the actual volume of the particular Sized ETT ( measured before intubation).
* The result obtained after this subtraction will be the volume of secretion or the volume of ETT that has been blocked.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anaesthesiologists (ASA) 1 and 2 adult Patients
2. Undergoing surgery for head and neck cancer
3. Requiring overnight endotracheal tube & breathing spontaneously

Exclusion Criteria:

1. Patients with major cardiac diseases( coronary artery disease, Valvular diseases)
2. Patients having gross chronic Obstructive Pulmonary Disease (COPD), bronchiectasis, cystic fibrosis.
3. Smokers(abstinence period less than 3 months)
4. Patient in drugs having sialogogue properties.
5. Patient on drugs having anti-sialogogue properties

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heated Humidifier Group | Mist Humidifier Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heated Humidifier Group | Mist Humidifier Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 20 | 42
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.57 (10.34) | 50.60 (11.60) | 49.58 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 22 | 21 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Extent of Blockade of Endotracheal Tube Assessed by Change in the Endotracheal Tube Volume
Description: The bevel end & Murphy's eye of the Endotracheal tube was sealed using sterile insulating tape so that it becomes water tight. The tube was gradually filled with measured amount of sterile fluid using small volume syringe to increase the accuracy of measurement. The amount of fluid it can hold was measured & noted
Time Frame: At baseline just before intubation and 24 hours from time of ICU admission
Measure: Mean (Standard Deviation); unit: percentage change of ET tube volume
Arm/Group | Heated Humidifier Group | Mist Humidifier Group
Number analyzed (Participants) | 30 | 30
percentage change of ET tube volume | 8.81 (6.35) | 14.08 (6.66)

2. Primary Outcome: Assess the Increase in Nurses Work Load
Description: Investigators will assess nursing workload by frequency of filling of humidifier chamber.
Time Frame: At baseline just before intubation and 24 hours from time of ICU admission
Population: The bevel end & Murphy's eye of the Endotracheal tube was sealed using sterile insulating tape so that it becomes water tight. The tube was gradually filled with measured amount of sterile fluid using small volume syringe to increase the accuracy of measurement. The amount of fluid it can hold was measured & noted
Measure: Mean (Standard Deviation); unit: time of refilling of nebuliser chamber
Arm/Group | Heated Humidifier Group | Mist Humidifier Group
Number analyzed (Participants) | 30 | 30
time of refilling of nebuliser chamber | 0.0 (0.0) | 3.5 (0.99)

ADVERSE EVENTS:
Arm/Group | Heated Humidifier Group | Mist Humidifier Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes